CLINICAL TRIAL: NCT01534897
Title: Re-differentiation of Radioiodine-Refractory BRAF V600E-mutant Papillary Thyroid Carcinoma With GSK2118436
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Lori J. Wirth, MD, Attending Physician, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-337
Record Dates: First submitted 2012-02-10; First posted 2012-02-17 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: Papillary Thyroid Carcinoma
Keywords: thyroid cancer; Tall cell PTC; Poorly differentiated thyroid carcinoma; metastatic
MeSH Terms: conditions — Thyroid Cancer, Papillary; Thyroid Neoplasms; Neoplasm Metastasis | interventions — dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GSK2118436 (Experimental): Intervention: GSK2118436 (dabrafenib) 150mg by mouth twice per day for 28 days, continued to day 42 if the Day 25 Iodine-131 scan shows new uptake. Patients with new Iodine-131 uptake on Day 25 who continue dabrafenib to day 42 receive a treatment dose (150 mCi) of Iodine-131 on Day 37.
  Interventions: Drug: GSK2118436

INTERVENTIONS:
Drug: GSK2118436 — 150mg twice per day orally for 28 days (42 days if Iodine-131 scan on Day 25 shows new uptake)
  Other Names: Dabrafenib

SUMMARY:
Radioactive iodine therapy is often part of the standard treatment for Papillary Thyroid Carcinoma (PTC) patients. However, in many patients, tumors develop a resistance or no longer respond to radioactive iodine therapy (iodine-refractory). Several lines of evidence suggest that blocking the BRAF gene may help to re-sensitize the tumors to radioactive iodine. BRAF is a protein that plays a central role in the growth and survival of cancer cells in some types of PTC. The investigational drug GSK2118436 may work by blocking the BRAF protein in cancer cells lines and tumors that have a mutated BRAF gene.

In this research study, the investigators are looking to see if GSK2118436 can re-sensitize iodine-refractory PTC to radioactive iodine therapy. The investigators are also looking at the safety of adding GSK2118436 to radioactive iodine therapy.

DETAILED DESCRIPTION:
You will take GSK2118436 capsules by mouth for 28 straight days. If your Day 28 whole body radioactive iodine scan demonstrates significant uptake of iodine, you will take GSK2118436 for an additional 14 days (Days 29-42). You will be given a drug diary to record when you take GSK2118436. This diary will also contain instructions on how to take GSK2118436.

Prior to Day 1

* Optional fine needle aspirate (pre-treatment) Day 1
* Vital signs
* Routine blood tests (2 tablespoons)
* Research blood sample for Circulating Tumor Cells (CTCs). (4 teaspoons of blood)
* Optional research blood sample for CTCs 4-6 hours after the first dose of GSK2118436

Day 2:

* Optional research blood sample for CTCs 4-6 hours after the first dose of GSK2118436 Day 3-5: Research blood sample for CTCs Days 8 and 15
* Vital signs
* Routine blood tests (2 tablespoons)
* Research blood sample for CTCs. (4 teaspoons of blood)
* Optional fine needle aspirate (Day 15 only) Low Iodine Diet: You will begin a low iodine diet on Day 15, in preparation for Day 23 when you will receive radioactive iodine (131I). The study team will provide you with instructions on this diet. The low iodine diet will be continued until the whole body scan is complete. For those participants who will receive a therapeutic dose of radioactive iodine on Day 37, the low iodine diet will be continued until the Day 42 whole body scan is complete.

Days 21 and 22: The drug thyrogen will be administered as in injection into your buttocks on Days 21 and 22 in preparation for your whole body radioactive iodine scan on Day 28. Thyrogen is used as a diagnostic tool to help determine the status of your cancer and is approved for use in thyroid cancer patients.

Day 23: To prepare for the whole body radioactive iodine scan, you will be asked to swallow a capsule of radioactive iodine which will be absorbed by any remaining thyroid cells in your body. Radioactive iodine is approved for use in thyroid cancer patients. You will then be asked to return for the scan on Day 28.You will be asked to sign a separate consent for the radioactive iodine.

Days 1-28:

* Optional repeat fine needle aspirate Day 28
* Whole body radioactive iodine scan to assess your thyroid cancer

If your Day 28 whole body radioactive iodine scan demonstrates significant uptake of iodine, you will have the following tests done within 24 hours:

* Vital signs
* Routine blood tests (2 tablespoons)
* Research blood sample for CTCs. (4 teaspoons of blood)
* An injection of a therapeutic dose of radioactive iodine will be administered. If your Day 28 whole body radioactive iodine scan does not demonstrate significant uptake of iodine, you will be removed from the research study. You will have a 3 month follow up appointment as outlined below.

If your Day 28 whole body radioactive iodine scan demonstrates significant uptake of iodine, you will continue treatment with GSK2118436 and have the following study visits:

Days 35 and 36: The drug thyrogen will be administered as in injection into your buttocks on Days 35 and 36 in preparation for your whole body radioactive iodine scan on Day 42.

Day 37: You will be given a therapeutic dose of radioactive iodine. You will be given a separate consent form to sign for your radioactive iodine treatment. You will then be asked to return for the whole body radioactive iodine scan on Day 42.

Day 39:

* Vital signs
* Routine blood tests (1 tablespoon)

Day 42:

* Whole body radioactive iodine scan
* Research blood sample for CTCs. (4 teaspoons of blood)

After the final dose of the study drug: All participants will have a follow up visit 3 months after you stop the study drug. You will have the following tests at this visit:

* Routine blood tests (2 tablespoons)
* Research blood sample for CTCs. (4 teaspoons of blood)
* An assessment of your tumor by CT scan or PET/CT scan of your neck, chest, abdomen and pelvis.
* Those participants who had a therapeutic dose of radioactive iodine on Day 37 will have a whole body radioactive iodine scan.
* Optional fine needle aspirate

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed papillary thyroid carcinoma, including its variants, such as tall cell PTC or poorly differentiated thyroid carcinoma, that is metastatic or unresectable AND harbors a BRAF V600E mutation
* Evaluable disease, as defined by at least one lesion that can be accurately measured in at least one dimension on CT scan or ultrasound, if present in the neck
* Radioiodine-refractory disease
* Life expectancy > 6 months
* Able to swallow and retain oral medication
* Normal organ and marrow function

Exclusion Criteria:

* Pregnant or breastfeeding
* Previous treatment with a specific BRAF or MEK inhibitor
* Receiving any other study agents
* Known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GSK2118436, bovine TSH, mannitol or iodine
* Active gastrointestinal disease or other condition that will interfere significantly with the absorption of drugs
* History of known glucose-6-phosphate dehyrogenase (G6PD) deficiency
* Corrected QT interval >/= 480 msecs; history of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within the past 24 weeks; Class II, III, or IV heart failure, abnormal cardiac valve morphology; or history of known cardiac arrhythmias
* Taking herbal remedies
* Subjects with significant symptoms from their thyroid cancer, or have a large burden of rapidly progressive iodine-refractory PTC who are in need of other systemic therapy, as judged by their treating physician
* Uncontrolled current illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension or psychiatric illness/social situations that would limit compliance with study requirements
* History of a different malignancy unless disease-free for at least 5 years and deemed to be at low risk for recurrence
* HIV-positive on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Rothenberg, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rothenberg SM, McFadden DG, Palmer EL, Daniels GH, Wirth LJ. Redifferentiation of iodine-refractory BRAF V600E-mutant metastatic papillary thyroid cancer with dabrafenib. Clin Cancer Res. 2015 Mar 1;21(5):1028-35. doi: 10.1158/1078-0432.CCR-14-2915. Epub 2014 Dec 30. PMID 25549723
- See also: pubmed url for article — http://www.ncbi.nlm.nih.gov/pubmed/25549723

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: July 2012-July 2013 Location: Massachusetts General Hospital Cancer Center Medical Clinic Number of patients recruited: 10 Recruitment goal: 10
Pre-assignment Details: All patients recruited were enrolled, and all patients completed the study.
Groups:
- GSK2118436: Note: This is a single arm feasibility study.
  Intervention: GSK2118436 (dabrafenib) 150mg by mouth twice per day for 28 days, continued to day 42 if the Day 25 Iodine-131 scan shows new uptake. Patients with new Iodine-131 uptake on Day 25 who continue dabrafenib to day 42 receive a treatment dose (150 mCi) of Iodine-131 on Day 37.
  GSK2118436: 150mg twice per day orally for 28 days (42 days if Iodine-131 scan on Day 25 shows new uptake)
Period: Overall Study
Arm/Group | GSK2118436
Started | 10
Day 25 Iodine-131 Scan | 10
Day 37 Iodine-131 Treatment | 6
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GSK2118436
Number analyzed (Participants) | 10
Age, Customized [Number; unit: participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10
Type of tumor [Count of Participants; unit: Participants]
  Classic papillary | 5
  Tall cell papillary | 4
  Clear cell papillary | 1
Prior radioiodine treatments per patient [Median (Full Range); unit: treatments] | 2 [1 to 4]
Prior surgeries per patient (not including initial thyroidectomy) [Median (Full Range); unit: surgeries] | 3 [0 to 6]
Prior external-beam radiotherapy [Number; unit: participants] | 3
Prior chemotherapy [Number; unit: participants] | 0
Prior targeted therapy [Number; unit: participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: Increased Radioiodine Uptake
Description: Number of patients with radioiodine-refractory metastatic BRAF V600E-mutant PTC who have increased radioiodine uptake in their disease sites while on dabrafenib. Radioiodine uptake is assessed by whole body scan and areas of interest are identified by nuclear medicine physicians.
Time Frame: 25 days after start of Dabrafenib (GSK2118436)
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2118436
Number analyzed (Participants) | 10
Participants | 6

2. Secondary Outcome: Safety Analysis as Number of Participants With Adverse Events
Description: To evaluate the safety and tolerability, as determined by adverse event and serious adverse event reporting, of GSK2118436 in combination with whole body iodine scans (all patients) and treatment doses of radioactive iodine (patients whose tumors demonstrate significant iodine uptake).
Time Frame: 2 years
Population: All patients completed dabrafenib without dose modification.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2118436
Number analyzed (Participants) | 10
Participants
  Experienced an Adverse Event | 10
  Experienced a Serious Adverse Event | 0
  Experienced a Grade 3, 4, or 5 Adverse Event | 0

3. Secondary Outcome: Clinical Benefit as Measured by Change in Tumor Size
Description: To evaluate clinical benefit as measured by objective response rate per modified RECIST 1.1, which assesses changes in size of measurable tumors. (per RECIST, a partial response (PR) = at least 30% decrease in size of tumor; progressive disease (PD) = at least 20% increase in size of tumor; stable disease (SD) = neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2118436
Number analyzed (Participants) | 10
Participants
  Stable Disease by RECIST | 7
  Progressive Disease by RECIST | 1
  Partial Response by RECIST | 2

4. Secondary Outcome: Number of Participants Who Complete the Study With Minimal Delays and no Dose Reductions
Description: To determine the feasibility of: (a) administering GSK2118436 for 28 days in patients with BRAF V600E-mutant PTC, prior to whole body iodine scanning (all patients); and (b) administering GSK2118436 for an additional 14 days, prior to administering treatment doses of radioactive iodine (patients whose tumors demonstrate significant iodine uptake after 28 days of treatment).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2118436
Number analyzed (Participants) | 10
Participants | 10

5. Secondary Outcome: Clinical Benefit as Measured by Change in Thyroglobulin Level
Description: To evaluate clinical benefit as measured by change in serum tumor marker, thyroglobulin. Rising thyroglobulin is generally indicative of tumor growth.
Time Frame: 3 months after radioiodine therapy
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2118436
Number analyzed (Participants) | 10
Participants
  decrease in serum thyroglobulin | 4
  increase in serum thryoglobulin | 6

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | GSK2118436
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2118436 (N=10)
Skin Changes (Skin and subcutaneous tissue disorders) | 8 (15)
Fatigue (General disorders) | 5 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 5 (8)
Palmar-Plantar Erythrodysethesias (Skin and subcutaneous tissue disorders) | 4 (4)
Headache (General disorders) | 3 (3)
Epistaxis (Blood and lymphatic system disorders) | 2 (2)
Creatinine Increase (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Weight loss (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No